CLINICAL TRIAL: NCT00002339
Title: An Open Multicenter Trial of Fluconazole Oral Suspension in the Treatment of Esophageal Candidiasis in Immunocompromised Patients
Brief Title: A Study of Fluconazole in the Treatment of Fungal Infections of the Throat in Patients With Weakened Immune Systems
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 120; R-0220
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Candidiasis, Esophageal; HIV Infections
Keywords: Esophagitis; Fluconazole; Acquired Immunodeficiency Syndrome; Candidiasis; Immunocompromised Host
MeSH Terms: conditions — Candidiasis; HIV Infections; Esophagitis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole

INTERVENTIONS:
Drug: Fluconazole

SUMMARY:
To determine the safety, toleration, and efficacy of fluconazole oral suspension in the treatment of esophageal candidiasis in immunocompromised patients, including those with AIDS.

DETAILED DESCRIPTION:
Patients receive fluconazole oral suspension for a minimum of 3 weeks and maximum of 8 weeks. Patients are evaluated weekly, and treatment continues for 2 weeks after resolution of symptoms. Endoscopic exams and possibly biopsies are performed at baseline and at the end of treatment. Patients undergo follow-up at 2 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* AIDS or other immunocompromising condition.
* Candidal esophagitis.
* Life expectancy of at least 2 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Evidence of non-candidal systemic fungal infection.
* Abnormalities that may preclude esophagoscopy or endoscopy.
* Unable to tolerate fluconazole.
* Unable to give informed consent.
* Enrollment in other experimental trials of approved or non-approved drugs or systemic compounds (unless approved by the Pfizer Clinical Monitor).
* Other condition that would make patient unsuitable for enrollment.

Concurrent Medication:

Excluded:

* Concomitant oral or topical antifungal agent.
* Other experimental medications.

Patients with the following prior condition are excluded:

History of allergy to imidazoles or azoles.

Prior Medication:

Excluded:

* Any oral or topical antifungal therapy within the past 3 days. Active use of illicit or illegal drugs.

Ages: 13 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Houston Veterans Administration Med Ctr, Houston, Texas

REFERENCES:
- [Background] Agresti MG, de Bernardis F, Mondello F, Bellocco R, Carosi GP, Caputo RM, Milazzo F, Chiodo F, Giannini V, Minoli L, et al. Clinical and mycological evaluation of fluconazole in the secondary prophylaxis of esophageal candidiasis in AIDS patients. An open, multicenter study. Eur J Epidemiol. 1994 Feb;10(1):17-22. doi: 10.1007/BF01717446. PMID 7957784